CLINICAL TRIAL: NCT00049933
Title: Hormone Replacement Therapy and Prothrombotic Variants
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Bruce Psaty, Professor, Medicine and Epidemiology, University of Washington
Other Study IDs: 20425; 5R01HL068639-04 (NIH)
Record Dates: First submitted 2002-11-14; First posted 2002-11-15 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Cerebrovascular Accident; Myocardial Infarction; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Stroke; Myocardial Infarction; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To examine in postmenopausal women the potential interactions of hormone replacement therapy with other blood clotting factors on the risk of cardiovascular diseases such as heart attack or stroke.

DETAILED DESCRIPTION:
BACKGROUND:

Estrogens are prothrombotic. Recently, the Heart and Estrogen/progestin Replacement Study (HERS), renewed interest in the adverse effects of hormone replacement therapy (HRT). In HERS, HRT was no better than placebo at preventing coronary events. In post hoc analyses, treatment was associated with early harm and late benefit. In an American Heart Association funded case-control study, a potential interaction was observed between HRT and the prothrombin G20210A variant on the risk of first myocardial infarction (MI) in post-menopausal women with hypertension.

DESIGN NARRATIVE:

The study has a case-control design. The Group Health Cooperative (GHC) computerized files will be used to identify postmenopausal women, aged 30 to 79 yrs, with incident myocardial infarction (MI) or stroke during 1/2000-12/2004. Population-based controls, sampled from the GHC enrollment files, will be frequency matched to cases by age, calendar year, and treated hypertension. Data collection will include medical-record review, telephone interview of consenting subjects, and venous-blood collection. Standard methods will be used to assay variant alleles. The GHC computerized pharmacy records will serve as the primary source of information about the use of HRT. Data analysis will involve restriction, stratification, and logistic regression. Case-control and case-only analyses are planned. There will be a total of 600 MI cases, 420 stroke cases and 1800 controls.

The primary purpose is to examine the potential interactions of hormone replacement therapy with other procoagulant variants on the risk of cardiovascular events. The main variants of interest are: (la) factor XIIIA Val34Leu; (ib) platelet glycoprotein (PGP) Jib Ile843Ser; (ic) PGP IIIa Leu33Pro; and (id) PGP Ia C807T. The secondary aims include the assessment of other drug-gene, risk-factor-gene or gene-gene interactions on risk: (2a) the interaction between PGP IIb Ser843, PGP lila Leu33Pro and PGP Ia C807T and traditional cardiovascular risk factors such as smoking and obesity on the risk of MI and stroke; (2b) the interaction between three coagulation factor XIII polymorphisms and PAl-1 4G/5G on the risk of stroke in women; and (2c) the interaction between aspirin use and glycoprotein IIIa Leu33Pro on the risk of MI and stroke.

ELIGIBILITY:
No eligibility criteria

Ages: 30 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2002-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Myocardial Infarction or Stroke | Retrospective

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Psaty, Study Chair — University of Washington

REFERENCES:
- [Background] Psaty BM, Lumley T, Furberg CD, Schellenbaum G, Pahor M, Alderman MH, Weiss NS. Health outcomes associated with various antihypertensive therapies used as first-line agents: a network meta-analysis. JAMA. 2003 May 21;289(19):2534-44. doi: 10.1001/jama.289.19.2534. PMID 12759325
- [Background] Rhoads CS, Psaty BM, Olson JL, Furberg CD. Medications and cardiovascular health in older adults: room for improvement in prevention and treatment. Am J Geriatr Cardiol. 2004 May-Jun;13(3):161-7. doi: 10.1111/j.1076-7460.2004.02124.x. No abstract available. PMID 15133419
- [Background] Smith NL, Heckbert SR, Lemaitre RN, Reiner AP, Lumley T, Weiss NS, Larson EB, Rosendaal FR, Psaty BM. Esterified estrogens and conjugated equine estrogens and the risk of venous thrombosis. JAMA. 2004 Oct 6;292(13):1581-7. doi: 10.1001/jama.292.13.1581. PMID 15467060
- [Background] Tirschwell DL, Smith NL, Heckbert SR, Lemaitre RN, Longstreth WT Jr, Psaty BM. Association of cholesterol with stroke risk varies in stroke subtypes and patient subgroups. Neurology. 2004 Nov 23;63(10):1868-75. doi: 10.1212/01.wnl.0000144282.42222.da. PMID 15557504
- [Derived] Altorki N, Wang X, Damman B, Jones DR, Wigle D, Port J, Conti M, Ashrafi AS, Liberman M, Landreneau R, Yasufuku K, Yang S, Mitchell JD, Keenan R, Bauer T, Miller D, Kozono D, Mentlick J, Vokes E, Stinchcombe TE. Recurrence of Non-Small Cell Lung Cancer With Visceral Pleural Invasion: A Secondary Analysis of a Randomized Clinical Trial. JAMA Oncol. 2024 Sep 1;10(9):1179-1186. doi: 10.1001/jamaoncol.2024.2491. PMID 39088196